CLINICAL TRIAL: NCT04874402
Title: Prepectoral vs Partial Subpectoral Two-Stage Implant-Based Breast Reconstruction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator left institution
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CASE1121
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Breast Reconstruction Following Mastectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prepectoral approach (Active Comparator): Immediately following mastectomy, participants will undergo prepectoral reconstruction approach. Intraoperative filling volume will be decided by the attending surgeon based on the pocket dimension and volume capabilities. Participants will be evaluated at 6 time points during the study.
  Interventions: Procedure: Prepectoral approach
- Partial subpectoral approach (Experimental): Immediately following mastectomy, participants will undergo partial subpectoral reconstruction approach. Intraoperative filling volume will be decided by the attending surgeon based on the pocket dimension and volume capabilities. Participants will be evaluated at 6 time points during the study.
  Interventions: Procedure: Partial Subpectoral approach

INTERVENTIONS:
Procedure: Prepectoral approach — Two sheets of contour, fenestrated ADM sutured together are trimmed in accordance with the measurement of the expander/implant and fixed to the pectoralis major muscle (superiorly, medially, and inferiorly) and serratus fascia (laterally), covering the entire anterior surface of the device
  Arms: Prepectoral approach
Procedure: Partial Subpectoral approach — The leading edge of the pectoral muscle is elevated and a subpectoral pocket is fashioned. The lower medial origin muscle fibers are released for anatomical expander seating. An ADM sling is sutured from the leading edge of the pectoralis muscle to the inframammary fold (over the expander) and laterally to close the expander pocket. In both groups, the size of the expander and the intraoperative filling volume will be decided by the attending surgeon based on the pocket dimension and volume capabilities.
  Arms: Partial subpectoral approach

SUMMARY:
The purpose of this study is to investigate the to analyze the patient satisfaction and complication rates under controlled conditions of the increasingly popular prepectoral technique for implant-based breast reconstruction.

DETAILED DESCRIPTION:
This is a single center, single-blinded, randomized clinical trial involving adult women undergoing two-stage implant-based breast reconstruction for either breast cancer or breast cancer risk reduction. The aim is to generate high quality evidence before establishing the prepectoral technique as routine care. A favorable safety and patient satisfaction profile will bring high quality evidence supporting the adoption of a technique that has shown similar complication rates while eliminating animation deformity and its associated pain and discomfort in retrospective and non-randomized studies.

The mastectomy flap perfusion will be assessed clinically and using SPY fluorescence imaging. Immediately following mastectomy, participants will be randomized to one of two treatment arms.

Group A will be composed of participants who will undergo prepectoral reconstruction with Acellular Dermal Matrix (ADM) by means of the anterior tenting technique. In this technique, two sheets of contour, fenestrated ADM sutured together are trimmed in accordance with the measurement of the expander/implant and fixed to the pectoralis major muscle covering the entire anterior surface of the device

Group B (current standard of care (SOC)) will be composed of participants who will undergo partial subpectoral reconstruction with ADM by means of the sling technique. In this technique the leading edge of the pectoral muscle is elevated and a subpectoral pocket is fashioned. The lower medial origin muscle fibers are released for anatomical expander seating. An ADM sling is sutured from the leading edge of the pectoralis muscle to the inframammary fold (over the expander) and laterally to close the expander pocket.

ELIGIBILITY:
Inclusion Criteria:

- Undergoing two-stage implant-based breast reconstruction for either breast cancer or breast cancer risk reduction

Exclusion Criteria:

* Active use of any tobacco products
* Uncontrolled diabetes defined by HbA1c greater than 7.5%
* Class II obesity or higher defined by a body mass index equal or greater than 35 kg/m2
* History of radiation to the affect breast or chest
* Immunocompromised patients
* Clinical evidence of significant mastectomy flap ischemia prior to the initiation of the reconstructive procedure

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction as measured by BREAST-Q-scores | Preoperatively
  Patient satisfaction will be assessed using BREAST-Q-scores. BREAST-Q is a patient-reported outcome instrument used to assess the outcomes of different breast surgeries among women. Modules selected will be "Psychosocial Well-Being, Physical Well-Being: Chest and Satisfaction with Breasts" within the Reconstruction (Preoperative) module and "Psychosocial Well-Being, Physical Well-Being: Chest, Satisfaction with Breasts and Satisfaction with Implants" within the Reconstruction (Postoperative) module
  For each BRESAT-Q scale, items are summed and transformed to a score with range from 0 to 100, and with greater values representing more satisfaction and higher levels of breast related quality of life.
  A two-sample T-test will be used to assess the changes in mean scores of satisfaction between two arms
Patient satisfaction as measured by BREAST-Q-scores | postoperative day 90 +/-30 days
  Patient satisfaction will be assessed using BREAST-Q-scores. BREAST-Q is a patient-reported outcome instrument used to assess the outcomes of different breast surgeries among women. Modules selected will be "Psychosocial Well-Being, Physical Well-Being: Chest and Satisfaction with Breasts" within the Reconstruction (Preoperative) module and "Psychosocial Well-Being, Physical Well-Being: Chest, Satisfaction with Breasts and Satisfaction with Implants" within the Reconstruction (Postoperative) module
  For each BRESAT-Q scale, items are summed and transformed to a score with range from 0 to 100, and with greater values representing more satisfaction and higher levels of breast related quality of life.
  A two-sample T-test will be used to assess the changes in mean scores of satisfaction between two arms

SECONDARY OUTCOMES:
Overall complication rates | Preoperatively
  Overall complication rates in both arms. Fisher's exact test will be performed to evaluate the differences in overall and specific complication rates between the two arms
Overall complication rates | Postoperative day 1
  Overall complication rates in both arms. Fisher's exact test will be performed to evaluate the differences in overall and specific complication rates between the two arms
Overall complication rates | Postoperative day 7 +/-7 days
  Overall complication rates in both arms. Fisher's exact test will be performed to evaluate the differences in overall and specific complication rates between the two arms
Overall complication rates | Postoperative day 14 +/-7 days
  Overall complication rates in both arms. Fisher's exact test will be performed to evaluate the differences in overall and specific complication rates between the two arms
Overall complication rates | postoperative day 21 +/-7 days
  Overall complication rates in both arms. Fisher's exact test will be performed to evaluate the differences in overall and specific complication rates between the two arms
Overall complication rates | postoperative day 90 +/-30 days
  Overall complication rates in both arms. Fisher's exact test will be performed to evaluate the differences in overall and specific complication rates between the two arms
Specific complication rates | Preoperatively
  Presence of seroma, hematoma, superficial and deep surgical site infection, wound dehiscence, skin necrosis, capsular contracture, rippling/visibility/palpability, and implant loss. Furthermore, the complications will be classified in major or minor based on the need for a surgical intervention to treat the complication or not, respectively.
  Fisher's exact test will be performed to evaluate the differences in overall and specific complication rates between the two arms
Specific complication rates | Postoperative day 1
  Presence of seroma, hematoma, superficial and deep surgical site infection, wound dehiscence, skin necrosis, capsular contracture, rippling/visibility/palpability, and implant loss. Furthermore, the complications will be classified in major or minor based on the need for a surgical intervention to treat the complication or not, respectively.
  Fisher's exact test will be performed to evaluate the differences in overall and specific complication rates between the two arms
Specific complication rates | Postoperative day 7 +/-7 days
  Presence of seroma, hematoma, superficial and deep surgical site infection, wound dehiscence, skin necrosis, capsular contracture, rippling/visibility/palpability, and implant loss. Furthermore, the complications will be classified in major or minor based on the need for a surgical intervention to treat the complication or not, respectively.
  Fisher's exact test will be performed to evaluate the differences in overall and specific complication rates between the two arms
Specific complication rates | Postoperative day 14 +/-7 days
  Presence of seroma, hematoma, superficial and deep surgical site infection, wound dehiscence, skin necrosis, capsular contracture, rippling/visibility/palpability, and implant loss. Furthermore, the complications will be classified in major or minor based on the need for a surgical intervention to treat the complication or not, respectively.
  Fisher's exact test will be performed to evaluate the differences in overall and specific complication rates between the two arms
Specific complication rates | postoperative day 21 +/-7 days
  Presence of seroma, hematoma, superficial and deep surgical site infection, wound dehiscence, skin necrosis, capsular contracture, rippling/visibility/palpability, and implant loss. Furthermore, the complications will be classified in major or minor based on the need for a surgical intervention to treat the complication or not, respectively.
  Fisher's exact test will be performed to evaluate the differences in overall and specific complication rates between the two arms
Postoperative pain intensity | Postoperative day 1
  Pain intensity evaluated using a visual analog scale. A mixed model with repeated measures will be conducted to analyze the differences in the postoperative pain at the immediate postoperative period and during the tissue expansion phase between the two arms
Postoperative pain intensity | Postoperative day 7 +/-7 days
  Pain intensity evaluated using a visual analog scale. A mixed model with repeated measures will be conducted to analyze the differences in the postoperative pain at the immediate postoperative period and during the tissue expansion phase between the two arms
Postoperative pain intensity | Postoperative day 14 +/-7 days
  Pain intensity evaluated using a visual analog scale. A mixed model with repeated measures will be conducted to analyze the differences in the postoperative pain at the immediate postoperative period and during the tissue expansion phase between the two arms
Postoperative pain intensity | postoperative day 21 +/-7 days
  Pain intensity evaluated using a visual analog scale. A mixed model with repeated measures will be conducted to analyze the differences in the postoperative pain at the immediate postoperative period and during the tissue expansion phase between the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Amir Ghaznavi, MD, Principal Investigator — Cleveland Clinic Florida, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Florida, Case Comprehensive Cancer Center, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD